CLINICAL TRIAL: NCT06848764
Title: A Randomized Double-Blind Trial Comparing Lidocaine and Dexmedetomidine Infusions for Intraoperative Bleeding in Patients Undergoing Functional Endoscopic Sinus Surgery
Brief Title: Lidocaine and Dexmedetomidine Infusions for Intraoperative Bleeding in Functional Endoscopic Sinus Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Monier Ahmed Youssef Eldemerdash, Lecturer of Anesthesia, Intensive care, and pain management Faculty of Medicine Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R42/2024/2025
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Lidocaine; Dexmedetomidine; Infusion; Intraoperative Bleeding; Functional Endoscopic Sinus Surgery
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Patients will receive lidocaine (1.5 mg/kg loading then 1mg/kg/h infusion) just after induction of anesthesia induction and continued until the end of the operation.
  Interventions: Drug: Lidocaine
- Dexmedetomidine group (Experimental): Patients will receive 1 μg/kg dexmedetomidine infusion over 10 min as a loading dose then 0.4-0.7 μg/kg/h just after induction of anesthesia induction and continued until the end of the operation.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Lidocaine — Patients will receive lidocaine (1.5 mg/kg loading then 1mg/kg/h infusion) just after induction of anesthesia induction and continued until the end of the operation.
  Arms: Lidocaine group
Drug: Dexmedetomidine — Patients will receive 1 μg/kg dexmedetomidine infusion over 10 min as a loading dose then 0.4-0.7 μg/kg/h just after induction of anesthesia induction and continued until the end of the operation.
  Arms: Dexmedetomidine group

SUMMARY:
This work aims to compare lidocaine and dexmedetomidine infusions for intraoperative bleeding in patients undergoing functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
Sinus surgery is one of the most prevalent surgeries on the ear, nose, and throat (ENT). It is mainly carried out through endoscopy and significantly improves the clinical symptoms of patients with rhinosinusitis. Safe conditions must be maintained for this surgery, and the major problem reported during functional endoscopic sinus surgery (FESS) under general anesthesia (GA) is impaired visibility due to excessive bleeding.

Dexmedetomidine is an α2-adrenoceptor agonist with sedative, anxiolytic, sympatholytic, analgesic-sparing effects and minimal depression of respiratory function. It is potent and highly selective for α2-receptors.

Lidocaine is an amino amide-type short-acting local anesthetic (LA). It has a short half-life and a favorable safety profile and is,, therefore,, the LA of choice for continuous IV administration.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* American Society of Anesthesiologists (ASA) physical status I - II.
* Scheduled for elective functional endoscopic sinus surgery.

Exclusion Criteria:

* Diabetes mellitus.
* Coagulation disorders.
* Kidney and liver dysfunction.
* Cerebrovascular disease.
* Cardiovascular problems.
* High blood pressure.
* Asthma.
* Chronic obstructive pulmonary disease (COPD).
* End organ damage.
* Psychosis.
* Taking antipsychotic drugs.
* Allergy to study drugs.
* Substance abuse.
* Taking beta blockers.
* Heart rate of < 55 beat/minute.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical field | Intraoperatively
  Surgical field will be assessed by Fromme et al. scale. (0-no bleeding, 1-slight bleeding, no suctioning of blood required, 2-slight bleeding occasional suctioning required, surgical field not threatened, 3-slight bleeding - frequent suctioning required. Bleeding threatens surgical field as few seconds after suction will be removed, 4-moderate bleeding - frequent suctioning required, bleeding threatens surgical field directly after suction will be removed, 5-severe bleeding - constant suctioning required, bleeding appeared faster than removed by suction. The surgical field severely threatened, and surgery not possible). The ideal category scale value will be determined to be ≤3.

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the VAS > 3 to be repeated after 30 min if pain persists until the Visual Analogue Scale (VAS)< 4. VAS will be assessed at post-anesthesia care unit (PACU), 2, 4, 6, 12, 18, and 24h postoperatively.
Heart rate | Till the end of surgery (Up to 4 hours)
  Heart rate will be recorded before induction, every 5 minutes for the first 20 minutes, then every 15 minutes until the end of the surgery.
Mean arterial pressure | Till the end of surgery (Up to 4 hours)
  Mean arterial pressure will be recorded before induction, every 5 minutes for the first 20 minutes, then every 15 minutes until the end of the surgery.
Time to the first request for the rescue analgesia. | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).
Degree of pain | 24 hours postoperatively
  The degree of pain will be assessed using the Visual Analogue Scale (VAS). (VAS 0 represents "no pain," while 10 represents "the worst pain imaginable.") VAS will be assessed at the post-anesthesia care unit (PACU), 2, 4, 6, 12, 18, and 24h postoperatively.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, upper airway obstruction, respiratory depression, emergence agitation, and postoperative awareness or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.